CLINICAL TRIAL: NCT06573684
Title: Differences In The Severity Of Diabetic Neuropathy Based On Electromyography In Type 2 Diabetes Mellitus Patients With And Without Comorbidities
Acronym: DISNEY-T2DM
Status: Completed | Type: Observational
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Maria Widiastuti, Prof, Professor, Universitas Diponegoro
Other Study IDs: Undip_Neuro
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Neuropathies
Keywords: Type II diabetic mellitus; Diabetic neuropathy; Electromyography
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type II Diabetic Mellitus without comorbidities: Patient who suffered diabetic neuropathy and history of type II diabetic mellitus without comorbidities
  Interventions: Diagnostic Test: Electromyography
- Type II Diabetic Mellitus with hypertension: Patient who suffered diabetic neuropathy and history of type II diabetic mellitus with hypertension
  Interventions: Diagnostic Test: Electromyography
- Type II Diabetic Mellitus with hypertension and dyslipidemia: Patient who suffered diabetic neuropathy and history of type II diabetic mellitus with hypertension and dyslipidemia
  Interventions: Diagnostic Test: Electromyography

INTERVENTIONS:
Diagnostic Test: Electromyography — All of groups will have assessment of electromyography result

SUMMARY:
The goal of this clinical trial is to learn the differences severity level of diabetic neuropathy based on electromyelography in type II diabetic patient with and without comorbidities. The main questions of this study:

1. What is the electromyography result in type II diabetic patient who: has no comorbidities, with hypertension, with hypertension and dyslipidemia?
2. Is there any differences in electromyography result in type II diabetic patient who: has no comorbidities, with hypertension, with hypertension and dyslipidemia?
3. Is there any association between distal latency with nerve conduction velocity in type II diabetic patient with and without comorbidities?
4. Is there any association between distal latency with amplitude in type II diabetic patient with and without comorbidities?
5. Is there any differences on diabetic neuropathy severity based on age, height, and A1C levels in type II diabetic patient with and without comorbidities?

Researchers will collect information based on hospital registry as secondary data of in type II diabetic patient with and without comorbidities. The data consist of demographic data, clinical presentation, laboratory, and electromyography were collected from hospital registry by reviewing medical record. Then, the data was analyzed by using IBM SPSS Statistics v26.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic neuropathy patient who classified as distal symmetrical polyneuropathy
* Diabetic neuropathy patient who has no comorbidities
* Diabetic neuropathy patient who has hypertension
* Diabetic neuropathy patient who has hypertension and dyslipidemia

Exclusion Criteria:

* Diabetic neuropathy patient with history of chemotherapy
* Diabetic neuropathy patient with history of hernia nucleus pulposus
* Diabetic neuropathy patient with history of CKD stage V or on routine dyalisis
* Missing data on medical record

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with type II diabetic mellitus who suffered diabetic neuropathy which diagnosed by using electromyography and fulfill the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Distal Latency | Electromyography examination was done approximately 1 year after clinical onset of neuropathy appear
  Distal latency defined as time between stimuli until deflection of Compound Muscle Action Potentials (CMAP) from baseline

SECONDARY OUTCOMES:
Nerve Conduction Velocity | Electromyography examination was done approximately 1 year after clinical onset of neuropathy appear
  Nerve Conduction Velocity defined as the measurement of axon conduction velocity by dividing space of nerve conduction with time needed
Amplitude | Electromyography examination was done approximately 1 year after clinical onset of neuropathy appear
  Amplitude define as the height of first negative deflection of Compound Muscle Action Potentials (CMAP) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Y, Xing P, Cai X, Luo D, Li R, Lloyd C, Sartorius N, Li M. Prevalence and Risk Factors for Diabetic Peripheral Neuropathy in Type 2 Diabetic Patients From 14 Countries: Estimates of the INTERPRET-DD Study. Front Public Health. 2020 Oct 20;8:534372. doi: 10.3389/fpubh.2020.534372. eCollection 2020. PMID 33194943
- [Background] England JD, Gronseth GS, Franklin G, Miller RG, Asbury AK, Carter GT, Cohen JA, Fisher MA, Howard JF, Kinsella LJ, Latov N, Lewis RA, Low PA, Sumner AJ; American Academy of Neurology; American Association of Electrodiagnostic Medicine; American Academy of Physical Medicine and Rehabilitation. Distal symmetric polyneuropathy: a definition for clinical research: report of the American Academy of Neurology, the American Association of Electrodiagnostic Medicine, and the American Academy of Physical Medicine and Rehabilitation. Neurology. 2005 Jan 25;64(2):199-207. doi: 10.1212/01.WNL.0000149522.32823.EA. PMID 15668414